CLINICAL TRIAL: NCT05213338
Title: Effect of Thermosensory Wear-documentation on Removable Orthodontic Appliance Compliance
Brief Title: Wear-documentation and Orthodontic Appliance Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: City of Vantaa (Other Government)
Responsible Party: Principal Investigator, Heidi Arponen, Principal investigator, DDS, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUS/3333/2021
Record Dates: First submitted 2022-01-03; First posted 2022-01-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Orthodontic Appliance Complication
Keywords: orthodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wear-documentation (Experimental): Theramon
  Interventions: Device: Wear-documentation microchip
- controls (No Intervention): No microchip

INTERVENTIONS:
Device: Wear-documentation microchip — Microchip embedded in the appliance
  Arms: wear-documentation

SUMMARY:
This randomized controlled trial aims to evaluate whether thermosensory wear-time documentation improves patient compliance of removable orthodontic appliances treated in a public health care clinic. The patients are children and adolescents.

DETAILED DESCRIPTION:
Qualitative subjective evaluation of appliance wear comfort and compliance is recorded, in addition to objective wear-time documentations.

ELIGIBILITY:
Inclusion Criteria:

* orthodontic treatment with removable appliances planned

Exclusion Criteria:

* non-compliance to participate in the study

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Treatment-time | through study completion, an average of 1 year
  months

SECONDARY OUTCOMES:
Patient satisfaction | through study completion, an average of 1 year
  qualitative self-evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Arponen, PhD, Principal Investigator — University of Helsinki
Locations (1):
- City of Vantaa, Vantaa, Finland

IPD SHARING:
Plan to Share IPD: No
Patient confidentiality prevents